CLINICAL TRIAL: NCT04464928
Title: Using Digital Media to Increase Population Knowledge of Urinary Incontinence Treatment Project
Brief Title: Pacific Northwest Female Urinary Incontinence Treatment Digital Awareness Project
Acronym: PNW-IP
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, W. Thomas Gregory, Professor of Obstetrics and Gynecology, Oregon Health and Science University
Other Study IDs: STUDY00020462
Record Dates: First submitted 2020-06-18; First posted 2020-07-09 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Urinary Incontinence
Keywords: female; advertising; urinary incontinence; social media; search engine; internet; quality of life; feasibility studies
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- User interests: Facebook advertisements arm
  Interventions: Other: Facebook Advertisements
- User characteristics: Google advertisements arm
  Interventions: Other: Google Advertisements

INTERVENTIONS:
Other: Facebook Advertisements — Counties will receive advertisements to VoicesForPFD.org's webpage on urinary incontinence on Facebook Ads when triggered by user characteristics indicating elevated risk of female urinary incontinence.
  Groups: User interests
Other: Google Advertisements — Counties will receive advertisements to VoicesForPFD.org's webpage on urinary incontinence on Google Ads when triggered by keywords relevant to female urinary incontinence.
  Groups: User characteristics

SUMMARY:
The investigators will compare whether advertisements on Google or Facebook are more effective to reach women in the Pacific Northwest about treatment options for urinary incontinence through the American Urogynecologic Society's patient education website, VoicesForPFD.org. The investigators hypothesize there is no difference in the overall population engagement between these two platforms due to anticipated higher reach through Facebook based on user characteristics but higher engagement through Google due to higher user interest on this platform.

DETAILED DESCRIPTION:
The investigators will conduct a comparative ecological study to compare effectiveness of two different targeted digital outreach platforms to engage women at risk for urinary incontinence in the Pacific Northwest. Counties in Oregon, Washington, Idaho will be randomized to receive advertisements for the American Urogynecologic Society's patient education website (domain VoicesForPFD.org) via either Google or Facebook. The investigators will use advertising campaigns developed specifically for this purpose. Through website analytics measuring advertisement clicks and census population data, the investigators will estimate utilization rates of the website for each county among the target population of middle-aged women to determine if one platform is more effective than the other for this topic and population.

ELIGIBILITY:
Inclusion Criteria:

- Internet user in Idaho, Oregon, or Washington states

Exclusion Criteria:

* Identified geographic location outside Idaho, Oregon, or Washington states
* Users identified by the advertising platforms as male.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Non-male users will be targeted based on their gender identification in each platform
Study Population: All internet users in all counties in Oregon, Washington, and Idaho will be eligible to see advertisements.
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Population website engagement | Through study completion, up to 4 months in duration from the start of advertising
  Number of website visits per capita through study advertisements.

SECONDARY OUTCOMES:
Impressions due to advertisements | Through study completion, up to 4 months in duration from the start of advertising
  Number of advertisement views per capita of the study advertisements.
Website users due to advertisements | Through study completion, up to 4 months in duration from the start of advertising
  Number of new users per capita coming to the VoicesForPFD.org website through study advertisements.

CONTACTS AND LOCATIONS:
Overall Officials: W Gregory, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be collected as part of the study.

REFERENCES:
- [Derived] Bennett AT, Boniface ER, Spiers A, Gregory WT, Cichowski SB. A Randomized Trial of Social Media Versus Search Engine Advertising to Increase Awareness of Treatments for Female Stress Urinary Incontinence. Female Pelvic Med Reconstr Surg. 2022 May 1;28(5):293-299. doi: 10.1097/SPV.0000000000001187. Epub 2022 Apr 15. PMID 35421015